CLINICAL TRIAL: NCT05583890
Title: A Case-control Study Comparing Glycaemic Control in Pancreatic Cancer Patients Versus Age Matched Healthy Individuals Using Continuous Glucose Monitors.
Brief Title: A Case-control Study Comparing Glycaemic Control in Pancreatic Cancer Patients vs Healthy Matched Individuals.
Acronym: PanCanCGM
Status: Completed | Type: Observational
Sponsor: Lancaster University (Other)
Collaborators: East Lancashire Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr. Chris Gaffney, Dr, Lancaster University
Other Study IDs: NHS REC no: 315235
Record Dates: First submitted 2022-10-11; First posted 2022-10-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
Keywords: Glycaemic control; Continuous glucose monitoring
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fitness Trackers; Diet Records; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy participants: Continuous glucose monitors will be fitted for 7 days, along with activity trackers and a food diary to monitor the impact of these factors on blood glucose concentrations. Participants will also complete questionnaires related to health inequalities and quality of life.
  Interventions: Device: Continuous glucose monitors; Device: Activity tracker; Behavioral: Food Diary; Behavioral: Questionnaires
- Pancreatic cancer patients undergoing chemotherapy: Continuous glucose monitors will be fitted for 7 days, along with activity trackers and a food diary to monitor the impact of these factors on blood glucose concentrations whilst they are undergoing chemotherapy. Participants will also complete questionnaires related to health inequalities and quality of life.
  Interventions: Device: Continuous glucose monitors; Device: Activity tracker; Behavioral: Food Diary; Behavioral: Questionnaires
- Pancreatic cancer patients not undergoing chemotherapy: Continuous glucose monitors will be fitted for 7 days, along with activity trackers and a food diary to monitor the impact of these factors on blood glucose concentrations. Participants will also complete questionnaires related to health inequalities and quality of life.
  Interventions: Device: Continuous glucose monitors; Device: Activity tracker; Behavioral: Food Diary; Behavioral: Questionnaires

INTERVENTIONS:
Device: Continuous glucose monitors — Participants will wear continuous glucose monitors for a 7 day period.
Device: Activity tracker — Participants will wear the activity tracker for a 7 day period.
Behavioral: Food Diary — Participants will complete a food diary of everything they eat for 7 days.
Behavioral: Questionnaires — Participants will complete FACT-Hep, DiPcare-Q and health inequality related questions.

SUMMARY:
The aim of this study is to continuously monitor blood glucose concentrations for a 7-day period in pancreatic cancer patients whilst undergoing their typical daily routines and to compare this to age matched healthy individuals. The investigators plan to carry out the study on a small subset of patients, up to 30 with pancreatic cancer (15 not undergoing chemotherapy and 15 undergoing chemotherapy) and 15 healthy individuals.

DETAILED DESCRIPTION:
The pancreas has two key functions related to digestion and metabolism. The first function of the pancreas is to produce exocrine enzymes which are released into the small intestine to help with the digestion of food. The second function is to produce endocrine hormones, such as insulin and glucagon, which help regulate glycaemic control. Impaired glucose metabolism and pancreatic cancer is temporally and pathogenically linked, with pancreatic tumours altering the secretion of key glucose regulatory hormones. Improved glucose regulation and lower glucose concentrations 3 months post-diagnosis of pancreatic ductal adenocarcinoma, a type of pancreatic cancer, has shown to increase overall survival.

The aim of this study is to continuously monitor blood glucose concentrations for a 7-day period in pancreatic cancer patients whilst undergoing their typical daily routines and to compare this to age matched healthy individuals. The comparison between healthy individuals and pancreatic cancer patients will investigate the severity of the difference between healthy glycaemic control and glycaemic control in those with pancreatic cancer. The comparison between pancreatic cancer patients undergoing chemotherapy and those not undergoing chemotherapy will help investigate the impact of chemotherapy on glycaemic control. This will help provide evidence as to what impact pancreatic cancer has on glycaemic control, whether continuous glucose monitors might be useful to regulate symptoms in patients, as a baseline to tailor an exercise intervention to regulate blood glucose concentrations and to investigate whether health inequalities impact glycaemic control.

The investigators plan to carry out the study on a small subset of patients, 30 with pancreatic cancer (15 undergoing chemotherapy and 15 not undergoing chemotherapy) and 15 healthy individuals.

ELIGIBILITY:
Pancreatic cancer patients

Inclusion Criteria:

* Aged 18-85
* Sex: male/female
* Radiological/tissue cancer diagnosis
* World Health Organisation performance status of 2 or below
* Patients with jaundice must have jaundice relieved before participating

Exclusion Criteria:

* Pregnancy
* Planned surgery within the 7 days of wearing the monitor
* Emergency surgery
* Part of any other trial with similar interventions
* Any musculoskeletal, cardiovascular, or neurological disorder that could put them at risk during the protocol.
* World Health Organisation performance status of above 2.
* Have diabetes at the point of diagnosis.

Healthy control group

Inclusion:

* Aged 18-85
* No serious underlying health conditions
* Age matched to pancreatic cancer patients

Exclusion:

* Take any medications which may alter blood glucose concentrations or insulin/glucagon concentrations, regular paracetamol intake during the study period, corticosteroids, thyroid hormones, or any anti-diabetes medication including insulin and oral hypoglycaemics.
* Pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients aged between 18 and 85 with a performance status of 2 and below. The patients must have jaundice relieved before participating and cannot have diabetes at the point of diagnosis.
  Healthy participants must be between 18-85 and age matched to the pancreatic cancer patients. The participants must not have any serious underlying health conditions or take any medications which may alter glycaemic control.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Glycaemic control | 7 day period
  Glycaemic control will be assessed by continuous glucose monitors for a 7-day period with activity trackers and food diaries used to further assess this control. The continuous glucose monitors takes readings every 5 minutes these readings will be averaged and area under the curve will be calculated.
Health inequalities | 7 day period
  Health inequalities, including household income, access to green space, main occupation, smoking habits, support system, ethnicity and religion assessed by specific questions and DipCare-Q questionnaires completed. Analyses determining the impact of inequalities on glyceamic control will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Gaffney, Principal Investigator — Lancaster University
Locations (2):
- United Kingdom (2):
  - Lancaster University, Lancaster, Lancashire
  - East Lancashire Hospitals Trust, Blackburn

IPD SHARING:
Plan to Share IPD: No